CLINICAL TRIAL: NCT06088004
Title: A Phase I/II Clinical Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics (PK/PD) and Preliminary Efficacy of ABO2011 Monotherapy or in Combination With Toripalimab in Patients With Advanced Solid Tumors
Brief Title: Phase Ⅰ/Ⅱ Clinical Study to Evaluate ABO2011 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Abogen Biosciences Co., Ltd. (Industry)
Collaborators: Abogen Biosciences (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABO2011-103
Record Dates: First submitted 2023-09-28; First posted 2023-10-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABO2011 (Experimental): Monotherapy
  Interventions: Drug: ABO2011 Injection
- ABO2011 and Toripalimab (Experimental): Combination therapy
  Interventions: Drug: ABO2011 Injection; Drug: Toripalimab

INTERVENTIONS:
Drug: ABO2011 Injection — Name of Active Ingredient: mRNA encoding human single-chain IL-12 protein; ABO2011 injection Route of administration: intratumoral injection
  Other Names: ABO2011; ABOD2011
Drug: Toripalimab — Anti-PD-1 antibody
  Arms: ABO2011 and Toripalimab

SUMMARY:
This is an open-label, single-arm, dose-escalation, and dose-expansion clinical study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of ABO2011 monotherapy or in combination with Toripalimab in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥18 years olde.
2. Ability to sign informed consent, including compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and this protocol.
3. Histopathology or cytology confirmed Advanced solid tumors;
4. Failed of previous systemic treatment or required treatment histories for selected tumor types;
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Expected survival greater than 12 weeks.
7. At least one superficial or deep lesion for intratumoral injection and biopsy.
8. Meet the required level of organ function.
9. Female patients are postmenopausal or, if women of childbearing potential, have a urine pregnancy or a blood pregnancy that is negative. At the same time, men of childbearing potential and women of childbearing potential voluntarily use effective contraception, including abstinence or effective contraception (e.g., intrauterine or implantable contraceptives, oral contraceptives, injectable or implantable contraceptives, extended-release local contraceptives, intrauterine devices [IUDs], condoms [males], diaphragms, cervical caps, etc.) from the time of signing the ICF until 120 days after the end of treatment.

Exclusion Criteria:

1. Other malignancies within the previous 5 years, with the exception of cured basal cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of breast, and carcinoma in situ of the cervix.
2. Central nervous system tumors or metastases with clinical symptoms or asymptomatic brain metastases requiring steroids control.
3. History of serious cardiac disease, e.g., New York Heart Association (NYHA) ≥ Grade 2 cardiac failure, history of transmural myocardial infarction, unstable angina, poorly controlled arrhythmia, myocardial infarction within 6 months prior to enrollment, or arrhythmias requiring antiarrhythmic therapy (β-blockers, calcium channel blockers, and digoxin are allowed). QTcF > 480 ms.
4. Poorly controlled clinical complications, including, but not limited to, uncontrolled hypertension with both antihypertensive agents Hypertension and hypoglycemic treatment not Controlled type 2 diabetes, poorly controlled pleural, ascites, or other serious diseases requiring systemic treatment.
5. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc.; type 1 diabetes mellitus, hypothyroidism controlled by replacement therapy only, and skin diseases that do not require whole body therapy (eg, vitiligo, psoriasis) may be included in the trial.
6. The subject carried: Known Human Immunodeficiency Virus (HIV); Active hepatitis B virus infection; Active hepatitis C virus infection.
7. Thrombotic disease or use of full-dose anticoagulant drugs within 6 months prior to screening.
8. Radiotherapy within 14 days prior to the first dose.
9. Live or live attenuated vaccines or other vaccines within 30 days prior to the first dose may be determined by the investigator's comprehensive assessment.
10. Major surgery within 28 days prior to the first dose or non-study-related minor surgery within 14 days prior to the first dose.
11. Immunosuppressants or other immunomodulatory medications are required within 4 weeks prior to the first dose, but physiologic doses of systemic steroids are allowed or topical. Topical use should not exceed the dose recommended in the package insert or have any signs of systemic exposure; or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation requiring the use of immunosuppressants or other immunomodulatory drugs.
12. Acute toxic effects of prior anticancer chemotherapy or immunotherapy have not been stable, or significant post-treatment toxicities have been observed.
13. Any systemic anti-tumor therapy with specific washout windows.
14. Presence of clinically significant pulmonary fibrosis or interstitial pneumonia.
15. Presence of active infections, including bacteria, fungi, viruses, and tuberculosis.
16. Active bleeding, including but not limited to gastrointestinal bleeding, hemoptysis, etc.
17. History of immediate severe allergic reactions prior to the first dose.
18. Other conditions that may increase the risk associated with the study drug, or affect the study compliance, which the investigator considers unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence and character of DLTs | monotherapy: 21 days after the first dose. Combination therapy: 28 days after the first dose]
Phase I: Incidence of Adverse Event (AE) | monotherapy: from informed consent until 28 days after the last administration. Combination therapy: from informed consent until 90 days after the last administration.
Phase I: Incidence of Serious Adverse Event (SAE) | monotherapy: from informed consent until 28 days after the last administration. Combination therapy: from informed consent until 90 days after the last administration.]
Phase I: Incidence of patients with clinically significant abnormal laboratory results | monotherapy: from the first dose until 28 days of last administration. Combination therapy: from informed consent until 90 days after the last administration.
Phase II: Objective response rates | Estimated to be from time of informed consent up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (5):
- China (5):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Guangxi Medical University Cancer Hospital, Nanning
  - Shanxi Cancer hospital, Shanxi
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen